CLINICAL TRIAL: NCT03993847
Title: CLassification of Axial SpondyloarthritiS Inception Cohort
Acronym: CLASSIC
Status: Completed | Type: Observational
Sponsor: Spondyloarthritis Research and Treatment Network (Network)
Collaborators: AbbVie (Industry); Amgen (Industry); Janssen Scientific Affairs, LLC (Industry); Eli Lilly and Company (Industry); Novartis Pharmaceuticals (Industry); Pfizer (Industry); UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: CLASSIC
Record Dates: First submitted 2019-06-12; First posted 2019-06-21 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Spondyloarthritis
Keywords: Spondyloarthritis; SPARTAN; ASAS; SpA; Undiagnosed Back Pain
MeSH Terms: conditions — Spondylarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Cohort of Undiagnosed Back Pain: All consecutive patients referred to a rheumatologist with current undiagnosed back pain of ≥3 months duration with onset ≤45 years of age will comprise the prospective cohort.
  This is a classification study; no intervention will be administered

SUMMARY:
A joint meeting of the ASAS (Assessment of Spondyloarthritis Internal Society) and SPARTAN (Spondyloarthritis Research and Treatment Network) executive boards recommended that the existing ASAS classification criteria for spondyloarthritis undergo further validation.

SPARTAN is in charge of conducting a a prospective study of a North American cohort of patients presenting with undiagnosed active chronic back pain to rheumatologists in the US and Canada, and one site in Mexico.

ASAS is in charge of conducting a similar study in Europe and other parts of the world.

DETAILED DESCRIPTION:
The overall study design will follow a similar format to that used to develop the ASAS axial SpA classification criteria. All consecutive patients referred to a rheumatologist with current undiagnosed back pain of ≥3 months duration with onset ≤45 years of age will comprise the prospective cohort. The sample size of 500 from North America (minimum of 300 from the US) and 500 from outside North America is aimed at ensuring that a sufficient number of patients will have axSpA and also permit the option to conduct 5-year follow up to determine predictive validity of the classification criteria. The clinical assessment data, including the history and physical examination, will be recorded by the rheumatologist in the electronic case report form (eCRF). This will be accessed through an online portal.

The rheumatologist will complete 5 global assessments to determine the presence/absence of axSpA. The first will be completed immediately after the first clinical assessment at the end of the patient encounter and will incorporate details of the history and physical exam. This is aimed at ascertaining which clinical features are considered most important in formulating the rheumatologist's opinion regarding the diagnosis of axSpA. The second will be conducted once the C-Reactive Protein (CRP), and HLA-B27 data are made available. The third will be completed after the pelvic radiograph has been reviewed by the rheumatologist. The fourth will be completed after the rheumatologist has reviewed the report of the pelvic MRI scan provided by the local radiologist. The fifth will be completed after central review of the anonymized radiograph and pelvic MRI scan and feedback to both the rheumatologist and radiologist. In ASAS centers outside North America, it may not be possible to have an assessment of each separate step as indicated if the rheumatologist already receives information on lab and imaging results in the referral later. In that circumstance, only global assessments 4 and 5 will be used as external standards. Patients will then be followed according to the discretion of the rheumatologist and appropriate standards of clinical practice. Patient contact information will be obtained and patient consent obtained through the informed consent to allow contact with the patient after 5 years of follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Undiagnosed back and/or buttock pain
2. Back, buttock or hip discomfort in the week before the study visit
3. Discomfort in the back, buttocks, or hips that has lasted at least three months.
4. First symptoms of pain when patient was ≤ 45 years of age:

Exclusion Criteria:

1. Patients with a known rheumatologist confirmed diagnosis of spondyloarthritis at the time of referral to the study-affiliated investigator.
2. Patients with a history of spinal trauma in the past 3 months.
3. Patients unable and/or unwilling to undergo MRI examination (embedded metallic fragments, pacemaker, joint replacement or similar hardware, too large (over 350 pounds unless their MRI can scan larger patients), claustrophobic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Undiagnosed back and/or buttock pain with onset ≤45 years and duration ≥ 3 months
Sampling Method: Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Physician diagnosis of axial spondyloarthritis at the final diagnostic evaluation. | 6 weeks
  Physician will answer Yes or No.

CONTACTS AND LOCATIONS:
Overall Officials: Walter P Maksymoywch, MD, Principal Investigator — Spondyloarthritis Research and Treatment Network
Locations (20):
- United States (15):
  - VA Long Beach Healthcare System, Long Beach, California
  - Sacramento VA Medical Center, Mather, California
  - UCSF Medical Center - Rheumatology Clinic, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia University, New York, New York
  - James J. Peters VAMC, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Dallas VA Medical Center VANTHCS, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Seattle Rheumatology Associates, Seattle, Washington
- Canada (3):
  - Artus Health Center, Vancouver, British Columbia
  - The Ottawa Hospital, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
- Mexico (2):
  - Centro de Estudios de Investigacion Basica y Clinica, SC, Guadalajara, Jalisco
  - CLIDITER, Mexico City, Mexico City

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Helliwell PS. 50 years of spondyloarthritis: a look back and a look ahead. Curr Opin Rheumatol. 2024 Jul 1;36(4):261-266. doi: 10.1097/BOR.0000000000001019. Epub 2024 Apr 24. PMID 38656252